CLINICAL TRIAL: NCT03266601
Title: Effect and Safety of Recombinant Human Interferon α-2b Spray on Herpangina in Pediatric Patients
Brief Title: Effect of Recombinant Human Interferon α-2b Spray on Herpangina
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: Tianjin Sinobioway Biomedicine Co.Ltd. (Unknown); Hunan Children's Hospital (Other Government); Children's Hospital of Chongqing Medical University (Other); Yuying Children's Hospital of Wenzhou Medical University (Other); Qilu Children's Hospital of Shandong University (Other); Children's Hospital of Kaifeng City (Unknown); Shenzhen Children's Hospital (Other Government); Zunyi Medical College (Other); Changhai Hospital (Other); Anhui Provincial Children's Hospital (Other)
Responsible Party: Principal Investigator, Hui Yu, Professor, Director, Children's Hospital of Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AFL-2015-2.0
Record Dates: First submitted 2017-08-10; First posted 2017-08-30 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Herpangina
Keywords: Aged 1-7 years old, within 72 hours of onset patients with herpangina
MeSH Terms: conditions — Herpangina | interventions — Ribavirin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recombinant Human Interferon α-2b Spray (Experimental)
  Interventions: Drug: Recombinant Human Interferon α-2b Spray
- Ribavirin (Active Comparator)
  Interventions: Drug: Ribavirin

INTERVENTIONS:
Drug: Recombinant Human Interferon α-2b Spray — Recombinant human interferon α-2b spray (trade name Jeferon, specifications: 1 million U/support, 10mL/support or 2 million U/support, 20mL/support, 2-8 ℃ dark storage and transportation), 1 million U/day, used for 3 days, observed to the 4th day (until the 96th hour).
  Arms: Recombinant Human Interferon α-2b Spray
Drug: Ribavirin — Ribavirin Spray, spray once every 4-5 hours, 1-2 times a spray, used for 3 days, observed to the 4th day(until the 96th hour ).
  Arms: Ribavirin

SUMMARY:
This is a multicenter, open，randomized controlled trial aiming to evaluate the effectiveness of recombinant human interferon α-2b spray compared with ribavirin treatment on pediatric patients with herpangina.

ELIGIBILITY:
Inclusion Criteria:

Subjects should meet all of the following:

1. meet the diagnostic criteria for pediatric herpangina;
2. ages 1-7 years, no limitation for gender;
3. within 72 hours of onset;
4. the main organs (heart, liver, kidney and lung) function normally;
5. follow up according to requirements and be hospitalized for observation;
6. the guardian is fully informed and signed informed consent.

Exclusion Criteria:

Subjects should be excluded if meet any of the following:

1. have allergy history of interferon;
2. heart failure, respiratory insufficiency,liver and kidney dysfunction or severe malnutrition and other serious disease, or immunodeficient;
3. children with epilepsy or other neurological disorders;
4. other pathogens exist at the same time;
5. the researchers believe that it is not appropriate to participate in this study.

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 668 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
The defervesce rate during treatment by 72 hours | Measure the body temperature every 4 hours from starting of treatment to the 96th hour.
  Body temperature returned to normal,and remain at least 24 hours.

SECONDARY OUTCOMES:
Abnormal blood routine | Before admission and 72th hours after treatment.
  White blood cell count, absolute neutrophil count, absolute lymphocyte count, platelet count, hemoglobin, the five indicators if one is abnormal, abnormal blood routine is defined as "1", if five indicators all are normal, abnormal blood routine is defined as "0".
The significant efficiency rate | From starting of treatment to the 48th hour.
  Within 48 hours treatment temperature returned to normal, oropharyngeal herpes and ulcers significantly improved and no new appeared, appetite significantly improved.
The effective rate | From starting of treatment to the 72th hour.
  Within 72 hours treatment temperature returned to normal, oropharyngeal herpes and ulcers improved and no new appeared, appetite improved.
The ineffective rate | From starting of treatment to the 96th hour.
  After medication 72 hours still fever, oropharyngeal herpes and ulcer without reducing or even increase, eating difficulty.
The total effective rate | From starting of treatment to the 96th hour.
  Total effective rate = efficiency rate + effective rate.
Total hospital stay | From starting of treatment to the 96th hour.
Appetite improvement | From starting of treatment to the 96th hour.
Myocardial enzymes and electrocardiogram | Before admission and 72th hours after treatment.
  Before admission myocardial enzymes and electrocardiogram were checked, then rechecked after 72 hours treatment if abnormal.
The condition of herpes and ulcers subside | Check the oral herpes or ulcers subsided every 24 hours from starting of treatment to the 72th hour.
  Clinical examination to check herpes subsided, ulcer wounds smaller, with or

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Fudan University, Shanghai, China